CLINICAL TRIAL: NCT04105959
Title: A Randomised, Single-Blind, Placebo-Controlled, Crossover Study to Investigate the Effects of RIST4721, a Novel CXCR2 Inhibitor, on the Inflammatory Response in Healthy Male Subjects Using a Standardized Blister Model
Brief Title: A Study to Investigate the Effects of RIST4721 on the Inflammatory Response in Healthy Male Subjects Using a Blister Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aristea Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RIST4721-102
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Inflammatory Response

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIST4721 300mg (Experimental): RIST4721 as once-daily 300mg oral solution for 6 days with a placebo crossover.
  Interventions: Drug: RIST4721; Drug: Placebo
- RIST4721 150mg (Experimental): RIST4721 as once-daily 150mg oral solution for 6 days with a placebo crossover.
  Interventions: Drug: RIST4721; Drug: Placebo

INTERVENTIONS:
Drug: RIST4721 — RIST4721 oral solution
Drug: Placebo — Placebo oral solution

SUMMARY:
A Randomised, Single-Blind, Placebo-Controlled, Crossover Study to Investigate the Effects of RIST4721, a Novel CXCR2 Inhibitor, on the Inflammatory Response in Healthy Male Subjects Using a Standardized Blister Model

ELIGIBILITY:
Inclusion Criteria:

* Subject is male, with Fitzpatrick skin types 1 to 3
* Subject is aged between 18 to 55 years, inclusive
* Subject has a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* Healthy as determined by a responsible physician, based on medical evaluation
* Must be willing to use birth control as indicated

Exclusion Criteria:

* Subject is known to have immune deficiency or is immunocompromised
* Subject has had a recent acute infection or chronic infection
* Subject has a known or suspected allergy or contraindications to cantharidin (blister induction method), RIST4721 or any component of the study drug
* Clinically relevant history of abnormal physical or mental health (including [but not limited to], neurological, psychiatric, endocrine, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Absolute neutrophil count in blister fluid at 24 hours post-blister formation compared to placebo | Blister formation to Hour 24
  Blister fluid will be harvested at 24, 30, and 36 hours post-blister formation and neutrophil count will be assessed at each time point and compared to placebo control
Absolute neutrophil count in blister fluid at 30 hours post-blister formation compared to placebo | Blister formation to Hour 30
  Blister fluid will be harvested at 24, 30, and 36 hours post-blister formation and neutrophil count will be assessed at each time point and compared to placebo control
Absolute neutrophil count in blister fluid at 36 hours post-blister formation compared to placebo | Blister formation to Hour 36
  Blister fluid will be harvested at 24, 30, and 36 hours post-blister formation and neutrophil count will be assessed at each time point and compared to placebo control

CONTACTS AND LOCATIONS:
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No